CLINICAL TRIAL: NCT00429468
Title: A Single-Centre, Double-Blind, Randomized, Placebo-Controlled, Phase 1 Study to Evaluate the Interaction Between Vicodin® CR and Ethanol in Healthy Male and Female Moderate Alcohol Drinkers
Brief Title: A Study to Evaluate the Interaction Between Vicodin® CR and Ethanol in Healthy Male and Female Moderate Alcohol Drinkers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: M06-835
Record Dates: First submitted 2007-01-29; First posted 2007-01-31 (Estimated); Last update posted 2007-10-26 (Estimated); Status verified 2007-10

CONDITIONS: Drug Interactions
MeSH Terms: interventions — Acetaminophen

INTERVENTIONS:
Drug: Vicodin® CR (extended-release hydrocodone/acetaminophen)

SUMMARY:
The purpose of this research study is to determine if varying strengths of ethanol affect the drug level and safety profile of Vicodin® CR.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ages 19 to 55
* If female, must be of non-child bearing potential or practicing birth control
* Current alcohol users who are classified as moderate drinkers (defined as 7-21 drinks per week)

Exclusion Criteria:

* Intolerance towards ethanol
* Is allergic to or has a serious reaction to hydrocodone, other opioids, or acetaminophen
* Significant GI narrowing or abnormality with a potential to inhibit GI motility or tablet transport
* History of seizures or convulsions, head injury or other intracranial lesions, or a pre-existing increase in intracranial pressure
* Has any clinically significant abnormalities on physical examination, ECG, or laboratory values
* Treatment with any investigational drug within 30 days of administration of study drug in the Treatment Phase

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25
Dates: Start 2007-01

PRIMARY OUTCOMES:
Standard pharmacokinetic assessments
statistical, clinical and laboratory procedures

CONTACTS AND LOCATIONS:
Overall Officials: Rita Jain, MD, Study Director — Abbott
Locations (1):
- Toronto, Ontario, Canada